CLINICAL TRIAL: NCT00225056
Title: Phase II Study of Capecitabine and Weekly Docetaxel Followed by Capecitabine Maintenance for Patients With Metastatic Breast Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to lack of accrual
Sponsor: Oncology Specialties, Alabama (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCIBRE02
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Capecitabine

INTERVENTIONS:
Drug: docetaxel and capecitabine

SUMMARY:
In this phase II study, we plan to evaluate the efficacy, safety and tolerability of weekly docetaxel and capecitabine on a 21-day cycle followed by maintenance single agent capecitabine for the treatment of metastatic breast cancer, Based on the efficacy and toxicity of the combination regimen dosages previously reviewed; weekly docetaxel 30mg/m2 on days 1 and 8 plus capecitabine 1600mg/m2 (800mg/m2 orally twice daily)on day 1 through 14 of each cycle will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* must have metastatic breast cancer
* must have cytologically or pathologically confirmed invasive ductal or lobular carcinoma
* must have measurable or evaluable disease
* ECOG of 0-1
* patients may have received 0, 1. or 2 prior treatments for metastatic breast cancer
* must have adequate organ function
* must be at least 19 years of age
* peripheral neuropathy less than or equal to grade 1
* must have voluntarily signed informed consent
* patients with brain metastases are eligible provided that other measurable disease exists and brain lesions are controlled

Exclusion Criteria:

* patients with other malignancies, except non melanoma of the skin, who have had any evidence of cancer within the last 5 years
* patients with psychiatric illness or other concurrent severe co-morbid medical condition that would preclude study completion
* known uncontrolled existing coagulopathy
* patients with a history of severe hypersensitivity reaction to docetaxel, medications formulated with polysorbate 80 or 5-fluorouracil
* use of other investigational agents in the last 28 days
* pregnant or lactating women
* patients who are known HIV positive
* patients with life expectancy of less than 3 months
* sexually active patients unwilling to practice reliable contraception during the study

Ages: 19 Years to 85 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 43
Dates: Start 2003-10; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Overall clinical benefit rate

SECONDARY OUTCOMES:
safety and tolerability
evaluate QOL
determine progression free survival
determine time to response and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: John M Waples, MD, Principal Investigator — Oncology Specialties, PC
Locations (1):
- Comprehensive Cancer Institute, Huntsville, Alabama, United States

REFERENCES:
- See also: Related Info — http://www.ccihsv.com